CLINICAL TRIAL: NCT04478045
Title: The Application of Point-of-care Ultrasonography in Differential Diagnosis of Shock in Emergency and Critical Care
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005121RINB
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-08

CONDITIONS: Shock; Ultrasonography; Differential Diagnosis; Emergencies; Critical Care
Keywords: Shock; Ultrasonography; Differential diagnosis; Emergency care; Critical care
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For the emergency physicians and critical care specialists, how to quickly recognize shock from diverse clinical features and immediately treat shock patients to prevent progression to irreversible organ dysfunction from initially reversible shock condition are important issues and challenges. In recent years, ultrasonography had been extensively used in clinical practice recently, and well-trained medical staffs can quickly and easily apply ultrasound to evaluate, examine, diagnose, and even treat the patients. The clinical application of point-of-care ultrasound can help the first-line physicians rapidly evaluate and diagnose the main symptoms and signs of the patients at bedside, and further initially stabilize and appropriately treat the patients subsequently. The aim of this program is to prospectively collection of the findings of point-of-care ultrasonography in shock patients at emergency room in NTUH. The clinical manifestations, and followed up the examinations, treatments, and prognosis will also be collected. The effect of bedside ultrasound on differential diagnosis and treatment of shock patients will be analyzed. The results of the current study can provide the base for further clinical trials and set up of shock team.

DETAILED DESCRIPTION:
Shock is defined as cellular and tissue hypoxia due to either reduced oxygen delivery, increased oxygen consumption, inadequate oxygen utilization, or a combination of these processes. According to the etiology about how it causes a decrease in blood flow to the cells and tissue, there are four types of shock naming cardiogenic shock, hypovolemic shock, obstructive shock, and distributive shock, respectively. The evaluation and management of shock patients is an extremely difficult challenge for the emergency physicians and critical care specialists. How to diagnose, classify, stabilize, and treat the shock patients quickly and in time are the arduous tasks. For the emergency physicians and critical care specialists, how to quickly recognize shock from diverse clinical features and immediately treat shock patients to prevent progression to irreversible organ dysfunction from initially reversible shock condition are important issues and challenges. In recent years, ultrasound instruments have gradually developed with higher radiographic quality and lower cost. Ultrasonography had been extensively used in clinical practice recently, and well-trained medical staffs can quickly and easily apply ultrasound to evaluate, examine, diagnose, and even treat the patients. The clinical application of point-of-care ultrasound can help the firstline physicians rapidly evaluate and diagnose the main symptoms and signs of the patients at bedside, and further initially stabilize and appropriately treat the patients subsequently. The aim of this program is to prospectively collection of the findings of point-of-care ultrasonography in shock patients at emergency room in NTUH. The clinical manifestations, and followed up the examinations, treatments, and prognosis will also be collected. The effect of bedside ultrasound on differential diagnosis and treatment of shock patients will be analyzed. The results of the current study can provide the base for further clinical trials and set up of shock team.

ELIGIBILITY:
Inclusion Criteria:

The shock patients in the emergency room at NTUH with one of the following conditions:

1. A clinician evaluated patients were with insufficient or improper tissue
2. Patients' systolic blood pressure < 90mmHg or mean arterial pressure < 65mmHg
3. Patients' laboratory data showed lactic acid > 2.2 mmol/L

Exclusion Criteria:

1. Age < 20 years
2. Pregnancy
3. Traumatic patients
4. Patients with DNR(Do Not Resuscitate) status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult, non-traumatic, non-DNR shock patients in the emergency room at NTUH are enrolled to our study. The point-of-care ultrasound in shock patients is performed by well-trained medical staffs.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The correlation between application of bedside ultrasound and differential diagnosis in shock patients | 6 month
  The effect of bedside ultrasound on differential diagnosis and treatment of shock patients.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, PhD, Study Director — National Taiwan University Medical College and Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan